CLINICAL TRIAL: NCT00244322
Title: LY450139: Tolerability and Biomarker Assessment in Subjects With Mild to Moderate Alzheimer's Disease
Brief Title: Effects of LY450139 Dihydrate on Subjects With Mild to Moderate Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 9097; H6L-MC-LFAJ
Record Dates: First submitted 2005-10-24; First posted 2005-10-26 (Estimated); Last update posted 2007-05-28 (Estimated); Status verified 2007-05

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

INTERVENTIONS:
Drug: LY450139 dihydrate
Drug: placebo

SUMMARY:
The purposes of this study are to determine:

* The safety of LY450139 dihydrate and any side effects that might be associated with it.
* How much LY450139 dihydrate should be given and how long it may be detected in blood.
* To determine if LY450139 dihydrate may have an effect on a protein found in blood, called A beta. This protein is studied in subjects with Alzheimer's disease.
* To collect and store samples from blood and spinal fluid for research related to Alzheimer's disease and similar (neurodegenerative) diseases or inflammation (irritation) that may provide information on how subjects respond to LY450139 or other medications.

Length of study: Approximately 29 weeks.

Number of office visits: 11 for most subjects: initial visit, every other week during 14 weeks of study drug treatment, and 2 follow-up visits.

At no cost, approximately 45 eligible participants will receive:

* Study medication
* Study-related diagnostic and laboratory evaluations

ELIGIBILITY:
Inclusion Criteria:

* At least 50 years of age and diagnosed with mild to moderate probable Alzheimer's disease
* Fluent in reading and speaking English and have a reliable study partner (caregiver) (someone who is in frequent contact and can make sure study medication is being taken correctly).
* If currently treated with certain drugs for Alzheimer's disease, doses must be the same for at least the last 2 months prior to starting study drug.

Exclusion Criteria:

* Cannot be currently using or require MAOI antidepressants (such as selegiline or Eldepryl(R)), antipsychotics, benzodiazepines, calcium channel blockers for heart disease, and propanolol.
* Cannot have a clinically significant and/or uncontrolled condition or other significant disease, including a condition requiring treatment with warfarin or heparin; or have had or currently have a peptic ulcer, reflux disease, or gastrointestinal (GI) bleeding.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45
Dates: Start 2005-10; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability

SECONDARY OUTCOMES:
Determine levels of peptides in blood and spinal fluid that might relate to Alzheimer's disease
Evaluate changes in thinking and memory
Evaluate changes in daily living activities
Determine levels of study drug in blood and spinal fluid

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (6):
- United States (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5hours, EST), or speak with your personal physician, La Jolla, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5hours, EST), or speak with your personal physician, Indianapolis, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5hours, EST), or speak with your personal physician, St Louis, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5hours, EST), or speak with your personal physician, Portland, Oregon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5hours, EST), or speak with your personal physician, Philadelphia, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5hours, EST), or speak with your personal physician, Seattle, Washington

REFERENCES:
- [Derived] Portelius E, Dean RA, Gustavsson MK, Andreasson U, Zetterberg H, Siemers E, Blennow K. A novel Abeta isoform pattern in CSF reflects gamma-secretase inhibition in Alzheimer disease. Alzheimers Res Ther. 2010 Mar 29;2(2):7. doi: 10.1186/alzrt30. PMID 20350302
- [Derived] Fleisher AS, Raman R, Siemers ER, Becerra L, Clark CM, Dean RA, Farlow MR, Galvin JE, Peskind ER, Quinn JF, Sherzai A, Sowell BB, Aisen PS, Thal LJ. Phase 2 safety trial targeting amyloid beta production with a gamma-secretase inhibitor in Alzheimer disease. Arch Neurol. 2008 Aug;65(8):1031-8. doi: 10.1001/archneur.65.8.1031. PMID 18695053
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com